CLINICAL TRIAL: NCT02429739
Title: Computerized Working Memory Training for Children With Dyslexia
Brief Title: Working Memory Training for Children With Dyslexia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sorlandet Hospital 2014/1057
Record Dates: First submitted 2015-04-24; First posted 2015-04-29 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Dyslexia
Keywords: Working Memory Training, computerized; Dyslexia; Reading fluency; Reading comprehension
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Working Memory Training (Experimental): Behavioral: Cogmed RM working memory training. After baseline assessment participants will be randomized to active training or treatment as usual (waiting). The active group will start immediately and will have 6 weeks to perform the 25 training sessions.
  Interventions: Behavioral: Working memory Training
- Passive control group (No Intervention): The control group will receive "treatment as usual" (Ordinary school days, special education if normally received).

INTERVENTIONS:
Behavioral: Working memory Training — The child will use the computer program at home under parental supervision for 25 sessions, each lasting 30 - 45 minutes and the family has 6 weeks to complete the training. Each session consist 8 different tasks presented by an animated robot. The tasks all require the child to hold information in working memory and to manipulate the information.
  Other name: Cogmed RoboMemo
  Arms: Working Memory Training

SUMMARY:
The main aim of this interventional study is to investigate whether the effects of computerized working memory training improves reading abilities for children, i.e. ages 9 - 16 years, diagnosed with dyslexia.

DETAILED DESCRIPTION:
Dyslexia is a specific learning difficulty which mainly affects the development of literacy and language related skills. It is characterized by difficulties with phonological processing, rapid naming, working memory, processing speed and the automatic development of skills that may not match up to an individual's other cognitive abilities. Phonological processing deficit is well established as one of the main causes of dyslexia. Working memory (WM) is today considered to be a cognitive system that strongly relates to a person's ability to think and learn. Over the last decade an increasing body of evidence indicates that WM deficits may cause particular problems for individuals with dyslexia. This is consistent with many of the every day problems reported by dyslexics and those around them. WM deficits are frequent in children with reading deficits. A major question is whether the WM impairment is secondary to phonological core deficit affecting the phonological loop only, or caused by an additional deficit involving central executive. Exploratory findings from fMRI studies indicates that impaired WM processes in dyslexia have a unique neuronal signature which may be associated with central executive processes. However there are conflicting findings and further studies are needed.

The children in the study, all diagnosed with dyslexia, will be divided into two subgroups (16/16 children). They are randomly allocated to either the adaptive training group or the treatment as usual control group after the baseline assessment. Both groups will meet for baseline testing and re-testing 4 weeks after completed training. Those that serve as non-trained controls will be offered to participate in training after completion of the study.

The intervention in this study aim to increase WM of children with dyslexia. We hypothesise that intensive computerized working memory training will improve reading fluency, speed and comprehension for children with dyslexia.

ELIGIBILITY:
Inclusion Criteria:

* Dyslexia

Exclusion Criteria:

* Mental retardation (IQ below 70)

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2014-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Reading fluency, comprehension and speed | Change from Baseline assessment to follow-up testing in 14 weeks
  LOGOS (http://www.logos-test.no) is a standardized Norwegian computerized test for reading processes. 6 subtest; reading fluency, reading comprehension, word recognition, phonological reading, orthographic reading, rapid naming of common objects

SECONDARY OUTCOMES:
Working Memory Capacity | Change from Baseline assessment to follow-up testing in 14 week
  WISC-IV: The sum of letter-number sequences and Digit Span, WMS-III Spatial Span, Språk 6-16 (Standardized Norwegian Screening-test for Language Impairment (Ottem &frost, 2011)Subtest: Sentence memory

OTHER OUTCOMES:
Executive function | Before and after training period of 5 weeks
  The ADHD Rating Scale-IV

CONTACTS AND LOCATIONS:
Overall Officials: Gro CC Lohaugen, Phd, Principal Investigator — Sorlandet Hospital HF
Locations (1):
- Sorlandet Hospital, Arendal, Aust-Agder, Norway

REFERENCES:
- [Background] Baddeley A. The episodic buffer: a new component of working memory? Trends Cogn Sci. 2000 Nov 1;4(11):417-423. doi: 10.1016/s1364-6613(00)01538-2. PMID 11058819
- [Background] Baddeley A. Working memory and language: an overview. J Commun Disord. 2003 May-Jun;36(3):189-208. doi: 10.1016/s0021-9924(03)00019-4. PMID 12742667
- [Background] Klingberg T. Training and plasticity of working memory. Trends Cogn Sci. 2010 Jul;14(7):317-24. doi: 10.1016/j.tics.2010.05.002. Epub 2010 Jun 16. PMID 20630350
- [Background] Klingberg, T (2012). Slik lærer hjernen. Oslo: Pax forlag
- [Result] Gathercole SE, Alloway TP. Practitioner review: short-term and working memory impairments in neurodevelopmental disorders: diagnosis and remedial support. J Child Psychol Psychiatry. 2006 Jan;47(1):4-15. doi: 10.1111/j.1469-7610.2005.01446.x. PMID 16405635
- [Result] Beneventi H, Tonnessen FE, Ersland L, Hugdahl K. Executive working memory processes in dyslexia: behavioral and fMRI evidence. Scand J Psychol. 2010 Jun 1;51(3):192-202. doi: 10.1111/j.1467-9450.2010.00808.x. Epub 2010 Mar 15. PMID 20338015
- [Result] Holmes J, Gathercole SE, Dunning DL. Adaptive training leads to sustained enhancement of poor working memory in children. Dev Sci. 2009 Jul;12(4):F9-15. doi: 10.1111/j.1467-7687.2009.00848.x. PMID 19635074
- [Result] Cogmed Working Memory Training (2012) Pearson assesment.no
- [Result] Hulme, C & Snowling, M.J.(2009) Developmental Disorders and Language Learning and Cognition, Chichester, WS.: Wiley - Blackwell
- [Result] Høien, T (2012) LOGOS; Teoribasert diagnostisering av lesevansker, Logometrica
- [Result] Ottem, E og Frost, J (2010) Språk 6-16 Screeningtest, Statped, Bredtvet kompetansesenter
- [Result] Swanson, H.L. (2006). Working memory and reading disabilities. I Alloway, T. & Gathercole, S (Red), Working Memory and Neurodevelopmental Disorders. (s. 59 - 88 9, Hove (UK): Psychology Press
- See also: Computerized Working Memory Training, RoboMemo — http://cogmed.com
- See also: Standardized Norwegian computerized test for reading processes — http://logometrica.no